CLINICAL TRIAL: NCT05843201
Title: Evaluation of Safety, Performance, and Usability of the AquaPass Device in Treatment of CHF Patients
Brief Title: AquaPass Device in Treatment of CHF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AquaPass Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQP-009
Record Dates: First submitted 2023-03-02; First posted 2023-05-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-11

CONDITIONS: Chronic Heart Failure; Edema; CHF
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients are hospitalized with chronic heart failure symptoms and fluid overloaded (Experimental): Phase 1: 'In Hospital' Phase: chronic heart failure (CHF) patients are enrolled in the study when admitted to the hospital with fluid overload.
  Study procedures performed, alongside diuretic therapy, in the hospital. Phase 2: 'At Home' Phase: Upon investigator's decision at discharge, the patients are enrolled in the second phase of the study for additional treatment sessions at home.
  Interventions: Device: The AquaPass System

INTERVENTIONS:
Device: The AquaPass System — The system is a non-invasive, multiple use device intended for use at the hospital, at the outpatient clinic settings or at home. The system administers warm, dry air around the patients' body in order to create environmental conditions that increase the patients' sweat rate. Throughout the treatment, fluids from the interstitial compartment are removed from the body by the eccrine sweat glands.

SUMMARY:
The AquaPass System is intended for enhancing fluid transfer through the skin, by increased sweat rate, in fluid overloaded patients.

This study will examine safety, performance and usability of the AquaPass device in two phases:

Phase 1: Hospitalization treatment. Phase 2: Home/outpatient clinic treatment

DETAILED DESCRIPTION:
The AquaPass System is intended for enhancing fluid transfer through the skin, by increased sweat rate, in fluid overloaded patients.

This study will examine safety, performance and usability of the AquaPass device in two phases:

Phase 1: Hospitalization treatment: This phase will begin when the patients are hospitalized with chronic heart failure symptoms and fluid overloaded and undergo sequential treatments. This phase will be conducted using a prospective case-control design, with measuring endpoint during hospitalization and follow-up (after discharge).

Phase 2: Home treatment: Upon investigator decision at discharge, patients will use Aqua-Pass device at home or at outpatient, after discharge, aiming to refine fluid management and prevent re-admission. This phase will require a separate Informed Consent Form (ICF) and will be conducted using a prospective single-group pre-post design.

* A multi-center, prospective, open label, one arm study.
* Chronic heart failure patients will be enrolled into the study when admitted to the hospital with fluid overload.
* During the in-hospitalization treatment phase, patients will undergo up to 5 procedures with the Aqua-Pass device between 3-8 hours.
* Following discharge and upon investigator decision, patients will sign a dedicated ICF and continue the Aqua-Pass treatments at home or in the outpatient clinic for up to 60 days, at a rate of 1-4 treatments per week.
* Follow up assessments, either during visit or over the phone, 7±2 days from the last procedure

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Subject was hospitalized for worsening of chronic heart failure with fluid overload.
3. Recruitment with expectation for at least 2 additional days in hospital.
4. Subject has composite congestion score ≥3.
5. Baseline systolic blood pressure ≥100.
6. Subject is capable of meeting the following study requirements:

   * Subject is taking a standing diuretic dose of ≥40 mg/day
   * For patients with BMI <30 kg/m2: baseline N-terminal pro b-type natriuretic peptide (NT-proBNP)>1,600 pg/ml
   * For patients with BMI >30 kg/m2: baseline N-terminal pro b-type natriuretic peptide (NT-proBNP) >800 pg/ml
   * For patients with rate-controlled persistent or permanent Atrial Fibrillation (AF): N-terminal pro b-type natriuretic peptide (NT-proBNP) >2,400 pg/ml.
7. Subject completes 2 hours of run-in acclimatization session as follows:

   * Put on the wearable and see if the patient fits inside it comfortably.
   * Turn on console and see if the patient feels well when the skin temperatures are at least 37°C.
   * Blood Pressure, Heart Rate, Core Temperature and have not changed, relative to baseline, by more than 20%.
   * Systolic BP does not drop below 90 mmHg in 2 consecutive measurements.

Exclusion Criteria:

1. Subject is enrolled to another clinical investigation that might interfere with this study.
2. Baseline systolic blood pressure <100 mm Hg
3. Subject considered to be in the acute worsening of the heart failure: Requiring ventilation, mechanical support or is clinically unstable requiring pressors, deterioration triggered by arrythmia, infection or other medical condition unrelated to fluid overload.
4. Subject has any known lower body skin problems (open wounds, ulcers)
5. Subject with severe peripheral arterial disease
6. Subject is pregnant or planning to become pregnant within the study period, or lactating mothers.
7. End-stage renal disease (eGFR<15 ml/min/1.73 m2) or requiring dialysis.
8. Inability or unwillingness to comply with the study requirements.
9. History of heart transplant or actively listed for heart transplant or Left Ventricular Assist Device (LVAD).
10. Implanted left ventricular assist device or implant anticipated <3 months.
11. Malignancy or other noncardiac condition limiting life expectancy to <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Rate of in-hospital procedures with fluid loss from sweat of >500 ml/session | In-Hospital Phase [2-10 days]
  The primary performance endpoint for the in-hospital phase is the amount of fluid loss from sweat per treatment procedure (~4h); the target rate of sweat production is >500 ml/session in the in-hospital phase.
Incidences of Device and treatment-related AEs and SAEs and symptomatic changes in vital signs | up to 70 days
  Symptomatic changes in vital signs including incidences of symptomatic hypotension and a decrease of more than 50% in eGFR compared to baseline

SECONDARY OUTCOMES:
Change in body weight | Up to 60 days
  To assess the effectiveness of the AquaPass System during the treatment phase patients will be assessed for their weight prior to the first treatment and after the last treatment
Change of diuretic therapy | Up to 60 days
  Documentation of changes in diuretics administration to assess safety and potential benefits with system use. (quantified by daily equivalent dose of furosemide).
Changes in NT-ProBNP levels | Up to 60 days
  Changes in NT-ProBNP levels to demonstrate the system's safety and performance
Rate of Hospitalizations or emergency visits for decompensated heart failure | Up to 60 days
  Documentation of CHF-related hospitalizations to assess safety and potential benefits with system use
Changes in Renal function | up to 60 days
  Changes in blood electrolytes that are correlated with worsening of renal function
Change of quality of life as assessed by the KCCQ-12 | Up to 60 days
  Patients will be asked to complete the KCCQ-12 Questionnaire to evaluate their QoL during the study and assess the potential effect of the treatment on their well-being

CONTACTS AND LOCATIONS:
Overall Officials: Doron Aronson, Prof., Principal Investigator — Rambam MC
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Rabin medical center, campus Belinson, Petah Tikva

IPD SHARING:
Plan to Share IPD: No